CLINICAL TRIAL: NCT03566017
Title: Open Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Pegunigalsidase Alfa (PRX-102) in Patients With Fabry Disease
Brief Title: Open Label Extension Study of 1 mg/kg Pegunigalsidase Alfa Every 2 Weeks in Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-06657AA1-04
Expanded Access: NCT04552691 (Approved for marketing)
Record Dates: First submitted 2018-05-24; First posted 2018-06-21 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease
Keywords: Glomerular filtration rate; Proteinuria; PRX-102; pegunigalsidase alfa; Fabry disease
MeSH Terms: conditions — Fabry Disease; Proteinuria

STUDY DESIGN:
Intervention Model Description: Open-label extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental open label (Experimental): pegunigalsidase alfa
  Interventions: Drug: pegunigalsidase alfa

INTERVENTIONS:
Drug: pegunigalsidase alfa — Recombinant human alpha galactosidase A
  Other Names: PRX-102

SUMMARY:
The objective of CLI-06657AA1-04 (formerly PB-102-F60) is to evaluate the long-term safety, tolerability, and efficacy parameters of 1 mg/kg pegunigalsidase alfa administered intravenously every other week in adult Fabry patients who have successfully completed studies PB-102-F03, PB-102-F20 or PB-102-F30.

DETAILED DESCRIPTION:
This is an open-label study. Patients will be enrolled to receive 1 mg/kg pegunigalsidase alfa as intravenous infusions every 2 weeks (±3 days). The duration of treatment is until pegunigalsidase alfa is commercially available to the patient, or at the discretion of the Sponsor. For the analysis, available efficacy and safety parameters will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of study PB-102-F20, PB-102-F03, or PB-102-F30
2. The patient signs informed consent
3. Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically acceptable method of contraception. These include combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal) supplemented with a barrier method (preferably male condom), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable) supplemented with a barrier method (preferably male condom), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, or sexual abstinence. Contraception should be used for 2 weeks after treatment termination.

Exclusion Criteria:

Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator, would interfere with patient compliance with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment-related adverse events | Throughout the study, 7 years
  CTCAE v4.03

SECONDARY OUTCOMES:
Kidney function 1 | Every 6 months throughout trial, 7 years
  Estimated glomerular filtration rate (eGFRCKD-EPI)
Cardiac assessment | Every 12 months to end of the study, 7 years
  Left Ventricular Mass Index (g/m2) by magnetic resonance imaging (MRI) and Echocardiograph, and exercise tolerance (Stress Test)
Biomarkers for Fabry disease | Every 12 months to end of the study, 7 years. For patients from PB-102-F20 at 3 and 6 months.
  plasma Lyso-Gb3 and Gb3
Record of pain medication use | Every two weeks for 7 years
  Frequency of pain medication use, or pre-infusion medication
Kidney function 2 | Every 6 months to the end of the study, 7 years
  Protein/Creatinine ratio, spot urine test (UPCR)
Pain assessment | Every 6 months up to the end of the study, 7 years
  short form Brief Pain Inventory (BPI)
Symptom assessment | Every 12 months up to the end of the study, 7 years
  Mainz Severity Score Index (MSSI)
Quality of life assessment | Every 6 months up to the end of the study, 7 years
  quality of life (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (15):
  - UAB Medicine, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of California Irvine Center, Orange, California
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Infusion Associates, Grand Rapids, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Renal Disease Research Institute, LLC - Dallas, Dallas, Texas
  - Institute of Metabolic Disease, Dallas, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - O+O Alpan LLC, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Royal Melbourne Hospital, Parkville, Victoria, Australia
- Capital District Health Authority, Halifax, Nova Scotia, Canada
- Vseobecna fakultni nemocnice v Praze, Prague, Czech Republic, Czechia
- Turku University Central Hospital, Turku, Finland
- Hospital Raymond-Poincaré, Garches, France
- Semmelweis Egyetem, Budapest, Hungary
- Azienda Ospedaliera Universitaria "Federico II", Napoli, Via Pansini, Italy
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Haukeland University Hospital Klinisk Forskningspost, Bergen, Norway
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- Hospital de Dia Quiron Zaragoza, Zaragoza, Spain
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Edgbaston, Birmingham
  - Salford Royal, Salford, Greater Manchester
  - Addenbrooke's Hospital, Cambridge
  - The Royal Free Hospital, London